CLINICAL TRIAL: NCT06949891
Title: Ketogenic Diet Therapy in Patients With Acromegaly
Acronym: KETOACRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Kirsten A Berk, RD, PhD, Senior Researcher, Assistant Professor, Department Internal Medicine - Dietetics (+31)107040567 k.berk@erasmusmc.nl Dr. Molewaterplein 40, 3015 GD Rotterdam Postbus 2040, 3000, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL8384107823
Record Dates: First submitted 2025-03-06; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Acromegaly Due to Pituitary Adenoma; Ketogenic Diet; Mediterranean Diet
MeSH Terms: conditions — Growth Hormone-Secreting Pituitary Adenoma | interventions — Diet, Ketogenic; Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- People with acromegaly following Ketogenic diet (Experimental): A eucaloric ketogenic diet (30-40 g carbohydrate per day) for 3 months, followed by a less strict ketogenic diet (50-60 g carbohydrate per day) for another 3 months.
  Interventions: Dietary Supplement: Ketogenic diet
- People with acromegaly following Mediterranean diet (Active Comparator): The control group will receive a eucaloric diet according to the national healthy food guidelines/Mediterranean diet.
  Interventions: Dietary Supplement: Mediterranean diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — A eucaloric ketogenic diet (30-40 g carbohydrate per day) for 3 months, followed by a less strict ketogenic diet (50-60 g carbohydrate per day) for another 3 months.
  Arms: People with acromegaly following Ketogenic diet
Dietary Supplement: Mediterranean diet — The control group will receive a eucaloric diet according to the national healthy food guidelines/Mediterranean diet.
  Arms: People with acromegaly following Mediterranean diet

SUMMARY:
Acromegaly is caused by a tumour located at the base of the brain in the pituitary gland that produces too much growth hormone (GH). Symptoms caused by the excess of GH, and consequently increased insulin like growth factor 1 (IGF-1), are disproportionate growth of body parts, fluid retention, snoring and excessive perspiration. The various metabolic changes that occur due to acromegaly increase the risk for insulin resistance, diabetes mellitus, arterial hypertension, sleep apnoea and thus an increased risk of cardiovascular disease if left untreated. The result is signs and symptoms, increased mortality, morbidity, and greatly reduced quality of life (QoL). Normalisation of GH and IGF-1 gives a normalisation of mortality, however morbidity and QoL do not (completely) normalise. After surgery, a somatostatin analogue is the primary medical treatment, however, normalisation occurs in only 40% of patients.

Recently, in a proof-of-principle study, the researchers showed that a 2-week ketogenic diet (low in carbohydrates) in patients with somatostatin analogues could significantly reduce IGF-1 values. Patients felt better and sometimes even needed less somatostatin analogues. This proof of concept led to the new hypothesis that acromegaly patients with somatostatin analogues should possibly be treated with a eucaloric low-carbohydrate ketogenic diet for a longer period of time to improve their biochemistry, symptoms and QoL. Additionally, this diet can make a significant contribution in the treatment of insulin resistance and glucose intolerance that often occur in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Diagnosis of acromegaly based on elevated GH and/or IGF-I levels due to a pituitary tumor
* IGF-I levels above 80% upper limit of the normal range (xULN)) on a stable medication dose for at least 4 months
* Written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Pegvisomant treatment
* Has undergone pituitary surgery or radiotherapy within 6 months prior to s study entry;
* It is anticipated that the patient will receive pituitary surgery or radiotherapy during the study;
* History or presence of epilepsy;
* Participation in a trail of an experimental drug or device within 30 days prior to screening;
* Has a mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
* Screening HbA1c > 6,5%;
* Use of antidiabetic medication other than Metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
IGF-1 | At baseline, 3 months and 6 months.
  Difference in IGF-1 (expressed as times the upper limit of the normal range (xULN) in nmol/L) between control and intervention group.

OTHER OUTCOMES:
Food intake | At baseline, 3 months and 6 months.
  Food intake (3-day food diary, via 'Eetmeter Voedingscentrum') in kcal, grams of carbohydrates, proteins, saturated fat and total fat, fibers and full-fledged diet (yes/no).
Quality of Life questionnaire | At baseline, 3 months and 6 months.
  Quality of Life questionnaire AcroQol (Acromegaly Quality of Life questionnaire); a 5 point likertscale assessing frequency of occurrence (always [1] to never [5]) or degree of agreement (completely agree [1] to completely disagree [5]) with the statements), which assesses physical and psychological aspects of quality of life in 22 questions.
Quality of Life questionnaire | At baseline, 3 months and 6 months.
  PASQ= QoL about symptoms (Patient-Assessed Acromegaly Symptom Questionnaire) and consists of 5 acromegaly-related symptoms (soft-tissue swelling, arthralgia, headache, excessive perspiration, and fatigue), which are measured on a scale of 0 to 8 points (a higher score indicating more severe symptoms), and a cumulative score (scale 0 to 40 points) can be calculated by adding the individual components )).
Qualtity of Life questionnaire | At baseline, 3 months and 6 months.
  D-KETOcheck questionnaire; consist of 11 questions of the ketogenic which are measured on a scale of 0-4 points (a higher score indicating stronger agreement to the ketogenic diet) for patients in arm of Ketogenic diet.
Serum parameters | At baseline, 3 months and 6 months.
  GH level in ug/l
Serum parameters | At baseline, 3 months and 6 months.
  IGF1 level in nmol/l
Serum Parameters | At baseline, 3 months and 6 months.
  Fasting plasma glucose in mmol/l
Serum parameters | At baseline, 3 months and 6 months.
  Fasting insulin in pmol/l
Serum parameters | At baseline, 3 months and 6 months.
  HbA1c in mmol/mol
Serum parameters | At baseline, 3 months and 6 months.
  Total cholesterol in mmol/l
Serum parameters | At baseline, 3 months and 6 months.
  HDL-cholesterol in mmol/l
Serum parameters | At baseline, 3 months and 6 months.
  LDL-cholesterol in mmol/l
Serum parameters | At baseline, 3 months and 6 months.
  Triglycerides in mmol/l
Serum parameters | At baseline, 3 months and 6 months.
  Free fatty acids in mmol/l
Serum parameters | At baseline, 3 months and 6 months.
  β-Hydroxybutyrate in mmol/l
Anthropometry | At baseline, 3 months and 6 months.
  Height in m
Anthropometry | At baseline, 3 months and 6 months.
  Weigth in kg
Anthropometry | At baseline, 3 months and 6 months.
  BMI in kg/m2
Anthropometry | At baseline, 3 months and 6 months.
  Fat mass in kg and in percent
Anthropometry | At baseline, 3 months and 6 months.
  Fat free mass (skeletal muscle mass) in kg
Anthropometry | At baseline, 3 months and 6 months.
  Body water in percent
Anthropometry | At baseline, 3 months and 6 months.
  Hand grip strength in kg
Anthropometry | At baseline, 3 months and 6 months.
  Resting energy expenditure in kcal/day.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol